CLINICAL TRIAL: NCT01929356
Title: The Influence of Chest Physiotherapy on Lung Function Parameters in Primary Ciliary Dyskinesia
Brief Title: Chest Physiotherapy and Lung Function in Primary Ciliary Dyskinesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZLMB001
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: lung function tests; chest physiotherapy
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chest physiotherapy (Experimental): session of 20 minutes chest physiotherapy with physiotherapist, use of airway clearance techniques, PEP (positive expiratory pressure) device
  Interventions: Procedure: Chest physiotherapy

INTERVENTIONS:
Procedure: Chest physiotherapy — 20 minutes of chest physiotherapy by physiotherapist

SUMMARY:
Primary ciliary dyskinesia (PCD) is a rare disease, caused by impairment of the motile cilia. Patients present with chronic upper and lower respiratory tract infections. The therapy is mainly supportive and based on that of cystic fibrosis. Chest physiotherapy is one of the cornerstones of the therapy, however the influence of chest physiotherapy on lung function (short term and long term) is not clear. For interpretation of longitudinal lung function data it is important to examine the short time effect of chest physiotherapy. We hypothesize that a session of chest physiotherapy improves lung function and that thus lung function tests must be performed in a standardized way.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is a rare disease, caused by congenital dysfunction of the motile cilia, located in the upper and lower respiratory tract, in the reproductive system and in the embryonal node. Ineffective ciliary beating results in disturbed mucociliary clearance, which is an important defense mechanism in the respiratory tract. It causes recurrent and chronic upper and lower respiratory tract infections, leading to reversible (mucus plugging) and irreversible lung damage (bronchiectasis, atelectasis, mucus plugging). Just like cystic fibrosis, it is characterized by obstructive lung disease, measured by spirometry.

Using Multiple Breath Washout measurements, it has been shown that peripheral airways disease is present in PCD. Probably, MBW parameters are already abnormal before forced expiratory volume in one second is abnormal.

The therapy for patients with PCD is mainly supportive: regular oral or intravenous antibiotics to treat airway infections and chest physiotherapy to actively increase mucociliary clearance. Chest physiotherapy has the objective to clear mucus from the lungs. Guidelines support the treatment of patients with PCD with chest physiotherapy. It is known that in patients with PCD, exercise has a more bronchodilating effect than the administration of salbutamol. However, no objective data describe the acute effect of chest physiotherapy on spirometry and MBW parameters. Moreover, short term effects of intervention on spirometry and MBW parameters can influence the interpretation of long-term evolution of these parameters.

In cystic fibrosis, one study has assessed the short-term influence of chest physiotherapy on lung function, measured by spirometry and MBW before and after chest physiotherapy. The authors found no significant influence of chest physiotherapy on spirometry parameters, nor on MBW parameters. Therefore, longitudinal interpretation can be performed irrespective of the timing of the lung function measurements. However, cystic fibrosis and PCD have a different pathophysiological mechanism with a more 'mechanical' disturbance of the mucociliary clearance in PCD, compared to a more 'viscous' disturbance of mucociliary clearance in CF. Therefore, the results in CF are not applicable to PCD. Even more, we hypothesize that chest physiotherapy will have a significant effect on lung function parameters (spirometry and MBW) in patients with PCD due to its external mechanical effect on mucus clearance.

ELIGIBILITY:
Inclusion Criteria:

* Primary ciliary dyskinesia
* able to perform spirometry and MBW (>6 years)

Exclusion Criteria:

* acute exacerbation

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Difference in FEV1 before and after treatment | 30 minutes
  Lung function will be performed before a session of chest physiotherapy, and repeated 30 minutes after a chest physiotherapy session of 20 minutes with airway clearance techniques and use of PEP mask

SECONDARY OUTCOMES:
Difference in LCI before and after chest physiotherapy | 30 minutes
  Multiple Breath Washout (MBW) will be performed before and 30 min after a session of chest physiotherapy. The difference in LCI (lung clearance index) will be used as secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Boon, MD, Principal Investigator — research fellow
Locations (1):
- University Hospital Gasthuisberg Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No